CLINICAL TRIAL: NCT03073187
Title: A Pilot Study to Improve Sleep Quality in Urban High School Students With Asthma
Brief Title: Sleep Quality in High School Students With Asthma
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jean-Marie Bruzzese, Professor of Applied Developmental Psychology (in Nursing), Columbia University
Other Study IDs: AAAQ9707 - I; 1R21HD086448-01A1 (NIH)
Record Dates: First submitted 2017-02-22; First posted 2017-03-08 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Asthma; Sleep; Asthma in Children
Keywords: Asthma; Sleep; Adolescents; Urban; Intervention; High school
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Students: Step 1 Interviews: 20 adolescents with uncontrolled asthma and poor sleep [10 from New York City (NYC); 10 from Rhode Island (RI)] will provide information regarding their asthma and sleep routines, and on what they would like to see in an intervention targeting co-morbid asthma and poor sleep.
- Caregivers: Step 1 Interviews: The caregivers of the 20 adolescents in this step [10 from NYC; 10 from RI] will be asked to provide information regarding their teenager's asthma and sleep routines, and on what they would like to see in an intervention targeting co-morbid asthma and poor sleep.
- Teachers: Step 2 Interviews: 4 high school teachers, 2 from NYC and 2 from RI, will review the developed intervention. They will provide their opinions about the appropriateness of the teaching methods and literacy level for adolescents.
- Students: Step 3 Focus Groups: 20 adolescents with uncontrolled asthma and poor sleep [10 from NYC; 10 from RI] will review the intervention providing feedback on its appropriateness and utility.
- Caregivers: Step 3 Focus Groups: The caregivers of the 20 adolescents in this step [10 from NYC; 10 from RI] will review the intervention providing feedback on its appropriateness and utility in small groups.

SUMMARY:
The overall goal of this project is to develop and to preliminarily validate a novel intervention to be delivered in the high school setting that integrates two evidence-based, school-based interventions for urban adolescents with proven efficacy: (1) Asthma Self-Management for Adolescents (ASMA), an intervention for adolescents with uncontrolled asthma and (2) the Sleep-Smart Program (Sleep-Smart), which focuses on sleep hygiene and behaviors in urban adolescents.

The aim for Phase I is to develop and integrate school-based interventions to improve asthma self-management and sleep hygiene in urban high school students via interviews.

The aims for Phase II are: (1) to evaluate the feasibility and acceptability of the intervention procedures; and (2) to assess the preliminary evidence of the effects of the intervention on improving sleep quality in urban high school students with persistent asthma over a 2-month follow-up period.

This record is for Phase I only.

DETAILED DESCRIPTION:
Sleep quality among adolescents is poor and asthma's impact is significant among adolescents. Asthma control is an important risk factor for poor sleep and poor academic performance. In addition, poor asthma control, poor sleep hygiene, and poor sleep quality are more likely in urban settings. Interventions to promote sleep quality by targeting both asthma control and sleep hygiene in this vulnerable population are lacking.

To adapt ASMA and Sleep-Smart, the investigators will use a 3-step iterative process that will consist of (1) interviewing high school students and their caregivers, (2) interviewing high school teachers and (3) conducting separate focus groups with students and caregivers. The investigators hypothesize that the intervention will be feasible and acceptable. This study is a multi-site trial and collaboration between Columbia University Medical Center and Rhode Island Hospital (RIH).

ELIGIBILITY:
ADOLESCENT-CAREGIVER DYADS (20 adolescents with persistent asthma and poor sleep, and their caregivers - 10 in Step 1 and 10 in Step 3)

Inclusion Criteria:

1. a prior asthma diagnosis in the prior 12 months;
2. use of prescribed asthma medications;
3. persistent asthma (defined as (i) daytime symptoms 3+ days a week, (ii) night awakenings 3+ nights per month, (iii) 2+ Emergency Department visits or (iv) 1+ hospitalization for asthma); and
4. sleep duration < 8 hours

Exclusion Criteria:

1. report of prior diagnosis of a sleep disorder, such as sleep disordered breathing, restless leg syndrome, periodic limb movement syndrome;
2. A Pediatric Sleep Questionnaire (PSQ) score of 0.33 or more, a well-validated measure of sleep disordered breathing risk;
3. active immunotherapy;
4. additional pulmonary disease; and
5. significant developmental delay and/or severe psychiatric or medical conditions that preclude completion of study procedures or confound analyses.

SCHOOL TEACHERS (4 high school teachers - 2 from New York and 2 from Rhode Island in Step 2)

Inclusion Criteria:

- Teach at the high school level.

Exclusion Criteria:

- Unwilling to participate in the study.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Families for Steps 1 and 3 will be identified through schools, clinics, and non-profit agencies that focus on asthma (e.g., American Lung Association). School principals, clinic directors, administrators and/or clinicians will distribute a flyer to families advertising the study, and families will be asked to call the researchers. In Rhode Island, families will also be recruited from their lab's database of past referrals and past research participants. Interested families will be screened for study eligibility by trained study staff.
  Each site will recruit two high school teachers for Step 2 from teachers known to the investigative team (convenient sample)
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Number of subjects successfully completing the interview | Up to 10 months
  Subjects will be interviewed regarding their preference and opinions about adapted curriculum.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Bruzzese, PhD, Principal Investigator — Columbia University; Daphne Koinis-Mitchell, PhD, Principal Investigator — Rhode Island Hospital
Locations (2):
- United States (2):
  - Columbia University, New York, New York
  - Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koinis-Mitchell D, Kopel SJ, Boergers J, McQuaid EL, Esteban CA, Seifer R, Fritz GK, Beltran AJ, Klein RB, LeBourgeois M. Good Sleep Health in Urban Children With Asthma: A Risk and Resilience Approach. J Pediatr Psychol. 2015 Oct;40(9):888-903. doi: 10.1093/jpepsy/jsv046. Epub 2015 May 18. PMID 25991645
- [Background] Vignau J, Bailly D, Duhamel A, Vervaecke P, Beuscart R, Collinet C. Epidemiologic study of sleep quality and troubles in French secondary school adolescents. J Adolesc Health. 1997 Nov;21(5):343-50. doi: 10.1016/S1054-139X(97)00109-2. PMID 9358298
- [Background] Meltzer LJ, Ullrich M, Szefler SJ. Sleep duration, sleep hygiene, and insomnia in adolescents with asthma. J Allergy Clin Immunol Pract. 2014 Sep-Oct;2(5):562-9. doi: 10.1016/j.jaip.2014.02.005. Epub 2014 Apr 13. PMID 25213049
- [Background] Wolfson AR, Carskadon MA. Understanding adolescents' sleep patterns and school performance: a critical appraisal. Sleep Med Rev. 2003 Dec;7(6):491-506. doi: 10.1016/s1087-0792(03)90003-7. PMID 15018092
- [Background] Wolfson AR, Carskadon MA. Sleep schedules and daytime functioning in adolescents. Child Dev. 1998 Aug;69(4):875-87. PMID 9768476
- [Background] Spilsbury JC, Storfer-Isser A, Drotar D, Rosen CL, Kirchner LH, Benham H, Redline S. Sleep behavior in an urban US sample of school-aged children. Arch Pediatr Adolesc Med. 2004 Oct;158(10):988-94. doi: 10.1001/archpedi.158.10.988. PMID 15466688
- [Background] Colrain IM, Baker FC. Changes in sleep as a function of adolescent development. Neuropsychol Rev. 2011 Mar;21(1):5-21. doi: 10.1007/s11065-010-9155-5. Epub 2011 Jan 12. PMID 21225346
- [Background] Dahl RE, Lewin DS. Pathways to adolescent health sleep regulation and behavior. J Adolesc Health. 2002 Dec;31(6 Suppl):175-84. doi: 10.1016/s1054-139x(02)00506-2. PMID 12470913
- [Background] Keyes KM, Maslowsky J, Hamilton A, Schulenberg J. The great sleep recession: changes in sleep duration among US adolescents, 1991-2012. Pediatrics. 2015 Mar;135(3):460-8. doi: 10.1542/peds.2014-2707. PMID 25687142
- [Background] Wong ML, Lau EY, Wan JH, Cheung SF, Hui CH, Mok DS. The interplay between sleep and mood in predicting academic functioning, physical health and psychological health: a longitudinal study. J Psychosom Res. 2013 Apr;74(4):271-7. doi: 10.1016/j.jpsychores.2012.08.014. Epub 2012 Sep 25. PMID 23497826
- [Background] Newacheck PW, Halfon N. Prevalence, impact, and trends in childhood disability due to asthma. Arch Pediatr Adolesc Med. 2000 Mar;154(3):287-93. doi: 10.1001/archpedi.154.3.287. PMID 10710030
- [Background] Worldwide variations in the prevalence of asthma symptoms: the International Study of Asthma and Allergies in Childhood (ISAAC). Eur Respir J. 1998 Aug;12(2):315-35. doi: 10.1183/09031936.98.12020315. PMID 9727780
- [Background] Centers for Disease Control and Prevention (CDC). Self-reported asthma among high school students--United States, 2003. MMWR Morb Mortal Wkly Rep. 2005 Aug 12;54(31):765-7. PMID 16094284
- [Background] Akinbami LJ, Moorman JE, Garbe PL, Sondik EJ. Status of childhood asthma in the United States, 1980-2007. Pediatrics. 2009 Mar;123 Suppl 3:S131-45. doi: 10.1542/peds.2008-2233C. PMID 19221156
- [Background] Pearce N, Ait-Khaled N, Beasley R, Mallol J, Keil U, Mitchell E, Robertson C; ISAAC Phase Three Study Group. Worldwide trends in the prevalence of asthma symptoms: phase III of the International Study of Asthma and Allergies in Childhood (ISAAC). Thorax. 2007 Sep;62(9):758-66. doi: 10.1136/thx.2006.070169. Epub 2007 May 15. PMID 17504817
- [Background] Akinbami LJ, Schoendorf KC. Trends in childhood asthma: prevalence, health care utilization, and mortality. Pediatrics. 2002 Aug;110(2 Pt 1):315-22. doi: 10.1542/peds.110.2.315. PMID 12165584
- [Background] Bloom B, Jones LI, Freeman G. Summary health statistics for U.S. children: National Health Interview Survey, 2012. Vital Health Stat 10. 2013 Dec;(258):1-81. PMID 24784481
- [Background] Bruzzese JM, Stepney C, Fiorino EK, Bornstein L, Wang J, Petkova E, Evans D. Asthma self-management is sub-optimal in urban Hispanic and African American/black early adolescents with uncontrolled persistent asthma. J Asthma. 2012 Feb;49(1):90-7. doi: 10.3109/02770903.2011.637595. Epub 2011 Dec 7. PMID 22149141
- [Background] Claudio L, Stingone JA, Godbold J. Prevalence of childhood asthma in urban communities: the impact of ethnicity and income. Ann Epidemiol. 2006 May;16(5):332-40. doi: 10.1016/j.annepidem.2005.06.046. Epub 2005 Oct 20. PMID 16242960
- [Background] Koinis-Mitchell D, McQuaid EL, Seifer R, Kopel SJ, Esteban C, Canino G, Garcia-Coll C, Klein R, Fritz GK. Multiple urban and asthma-related risks and their association with asthma morbidity in children. J Pediatr Psychol. 2007 Jun;32(5):582-95. doi: 10.1093/jpepsy/jsl050. Epub 2007 Jan 11. PMID 17218338
- [Background] Wright RJ. Further evidence that the wealthier are healthier: negative life events and asthma-specific quality of life. Thorax. 2007 Feb;62(2):106-8. doi: 10.1136/thx.2006.067926. PMID 17287304
- [Background] Williams DR, Sternthal M, Wright RJ. Social determinants: taking the social context of asthma seriously. Pediatrics. 2009 Mar;123 Suppl 3(Suppl 3):S174-84. doi: 10.1542/peds.2008-2233H. PMID 19221161
- [Background] Clark NM, Brown R, Joseph CL, Anderson EW, Liu M, Valerio M, Gong M. Issues in identifying asthma and estimating prevalence in an urban school population. J Clin Epidemiol. 2002 Sep;55(9):870-81. doi: 10.1016/s0895-4356(02)00451-1. PMID 12393074
- [Background] Koinis-Mitchell D, McQuaid EL, Kopel SJ, Esteban CA, Ortega AN, Seifer R, Garcia-Coll C, Klein R, Cespedes E, Canino G, Fritz GK. Cultural-related, contextual, and asthma-specific risks associated with asthma morbidity in urban children. J Clin Psychol Med Settings. 2010 Mar;17(1):38-48. doi: 10.1007/s10880-009-9178-3. PMID 20157798
- [Background] McLaughlin Crabtree V, Beal Korhonen J, Montgomery-Downs HE, Faye Jones V, O'Brien LM, Gozal D. Cultural influences on the bedtime behaviors of young children. Sleep Med. 2005 Jul;6(4):319-24. doi: 10.1016/j.sleep.2005.02.001. Epub 2005 Apr 1. PMID 15978515
- [Background] Redline S, Tishler PV, Schluchter M, Aylor J, Clark K, Graham G. Risk factors for sleep-disordered breathing in children. Associations with obesity, race, and respiratory problems. Am J Respir Crit Care Med. 1999 May;159(5 Pt 1):1527-32. doi: 10.1164/ajrccm.159.5.9809079. PMID 10228121
- [Background] Rosen CL, Palermo TM, Larkin EK, Redline S. Health-related quality of life and sleep-disordered breathing in children. Sleep. 2002 Sep 15;25(6):657-66. PMID 12224844
- [Background] Spilsbury JC, Storfer-Isser A, Kirchner HL, Nelson L, Rosen CL, Drotar D, Redline S. Neighborhood disadvantage as a risk factor for pediatric obstructive sleep apnea. J Pediatr. 2006 Sep;149(3):342-7. doi: 10.1016/j.jpeds.2006.04.061. PMID 16939744
- [Background] Boergers J, Koinis-Mitchell D. Sleep and culture in children with medical conditions. J Pediatr Psychol. 2010 Oct;35(9):915-26. doi: 10.1093/jpepsy/jsq016. Epub 2010 Mar 23. PMID 20332222
- [Background] Koinis-Mitchell D, Kopel SJ, Boergers J, Ramos K, LeBourgeois M, McQuaid EL, Esteban CA, Seifer R, Fritz GK, Klein R. Asthma, allergic rhinitis, and sleep problems in urban children. J Clin Sleep Med. 2015 Jan 15;11(2):101-10. doi: 10.5664/jcsm.4450. PMID 25515273
- [Background] Bruzzese JM, Bonner S, Vincent EJ, Sheares BJ, Mellins RB, Levison MJ, Wiesemann S, Du Y, Zimmerman BJ, Evans D. Asthma education: the adolescent experience. Patient Educ Couns. 2004 Dec;55(3):396-406. doi: 10.1016/j.pec.2003.04.009. PMID 15582346
- [Background] Bruzzese JM, Sheares BJ, Vincent EJ, Du Y, Sadeghi H, Levison MJ, Mellins RB, Evans D. Effects of a school-based intervention for urban adolescents with asthma. A controlled trial. Am J Respir Crit Care Med. 2011 Apr 15;183(8):998-1006. doi: 10.1164/rccm.201003-0429OC. Epub 2010 Dec 7. PMID 21139088
- [Background] Wolfson AR, Harkins E, Johnson M, Marco C. Effects of the Young Adolescent Sleep Smart Program on sleep hygiene practices, sleep health efficacy, and behavioral well-being. Sleep Health. 2015 Sep;1(3):197-204. doi: 10.1016/j.sleh.2015.07.002. Epub 2015 Aug 13. PMID 29073440